CLINICAL TRIAL: NCT00532311
Title: A Double-Blind, Randomized Study to Evaluate the Efficacy and Safety of Lapaquistat Acetate 50 mg or Placebo When Co-administered With Statins in Subjects With Hypercholesterolemia, With an Optional Open-Label Extension
Brief Title: Efficacy of Lapaquistat Acetate Co-Administered With Statins in Subjects With Hypercholesterolemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Overall profile of the compound does not offer significant clinical advantage to patients over currently available lipid lowering agents
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-475_307; U1111-1122-8479 (Registry Identifier: WHO)
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia; Drug Therapy
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid; Atorvastatin; Simvastatin; Rosuvastatin Calcium; Pravastatin; Fluvastatin; Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapaquistat Acetate 50 mg QD (Experimental): (and stable statin therapy)
  Interventions: Drug: Lapaquistat acetate and stable statin therapy
- Stable statin therapy (Active Comparator)
  Interventions: Drug: Stable statin therapy

INTERVENTIONS:
Drug: Lapaquistat acetate and stable statin therapy — Lapaquistat acetate 50 mg, tablets, orally, once daily and stable statin therapy for up to 12 weeks.
  Other Names: TAK-475; Lipitor; Zocor; Crestor; Pravachol; Lescol; Mevacor
  Arms: Lapaquistat Acetate 50 mg QD
Drug: Stable statin therapy — Lapaquistat acetate placebo-matching tablets, orally, once daily and stable statin therapy for up to 12 weeks.
  Other Names: Lipitor; Zocor; Crestor; Pravachol; Lescol; Mevacor
  Arms: Stable statin therapy

SUMMARY:
The purpose of the study is to determine the efficacy of lapaquistat acetate, once daily (QD), taken with statins on cholesterol levels in subjects with hypercholesterolemia

DETAILED DESCRIPTION:
Dyslipidemias are a group of metabolic disorders produced by raised concentrations of lipoproteins, especially low-density lipoprotein cholesterol, which is the lipoprotein that transports endogenous cholesterol from the liver to the peripheral tissues. Increased cholesterol and triglycerides levels lead to an increased risk of arteriosclerosis, which is the underlying cause of heart attack, strokes and peripheral vascular disease.

Despite changes in lifestyle and the availability of potent lipid-lowering agents, cardiovascular disease continues to be the major cause of death in Western Europe and North America. Serum cholesterol levels exceeding 5 mmol/L (193 mg/dL) are common in adults in Britain and much of Europe, the United States, Australia and New Zealand.

This study will evaluate the efficacy and safety of lapaquistat acetate taken with either torvastatin, simvastatin, rosuvastatin, pravastatin, fluvastatin or lovastatin (stable statin therapy) in subjects with hypercholesterolemia. Total participation time in this study is expected to be up to 12 weeks, with an optional, 48-week, open-label extension period for participants who qualify.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who are sexually active must agree to use adequate contraception from screening throughout the duration of the study and for 30 days following the last dose.
* Has been on a stable dose of statin for at least 3 months prior to Screening. Participants enrolled in Canada, Latin America, and South Africa must be on the maximum approved dose of statin (atorvastatin 80 mg, simvastatin 80 mg, rosuvastatin 40 mg, pravastatin 80 mg, fluvastatin 80 mg, or lovastatin 80 mg).
* Prior to Randomization, the participant has a mean low density lipoprotein cholesterol level greater than or equal to 100 mg/dL and less than or equal to 190 mg/dL for 2 consecutive samples.
* Prior to Randomization, the subject has mean triglyceride level greater than or equal to 400 mg/dL for 2 consecutive samples.
* Is willing and able to comply with the recommended, standardized diet.

Exclusion Criteria:

* Has an nine aminotransferase or aspartate aminotransferase level greater than 1.5 times the upper limit of normal, identified during screening.
* Has a serum creatinine greater than 133 mmol/L, identified during screening.
* Has a creatine kinase greater than 3 times the upper limit of normal, identified during screening.
* Has active liver disease or jaundice.
* Has taken any bile acid sequestrants [eg, cholestyramine], and intestinal cholesterol uptake inhibitors [eg, ezetimibe]) from 30 days before Screening until study completion or any fibrates for 6 weeks before Visit 1.
* Has a previous history of cancer that has been in remission for less than 5 years prior to the first dose of study medication.
* Has an endocrine disorder, such as Cushing's syndrome, hyperthyroidism, or inappropriately treated hypothyroidism affecting lipid metabolism.
* Has a history of myocardial infarction, angina pectoris, unstable angina, transient ischemic attacks, cerebrovascular accident, peripheral vascular disease, abdominal aortic aneurysm, coronary angioplasty, coronary or peripheral arterial surgery, or multiple risk factors that confer a 10-year risk for cardiovascular heart disease greater than 20% based on Framingham risk scoring.
* Has a positive hepatitis B surface antigen or hepatitis C virus antibody test, as determined by medical history.
* Has a positive human immunodeficiency virus status or is taking antiretroviral medications, as determined by medical history and/or subject's verbal report.
* Has received any investigational medication 30 days prior to screening, (for drugs with a long half-life, within a period of less than 5 times the drug's half-life) or is participating in an investigational study.
* Has received lapaquistat acetate in a previous clinical study or as a therapeutic agent.
* Has a history or presence of clinically significant food allergy that would prevent adherence to the specialized diet.
* Has a known heterozygous or homozygous familial hypercholesterolemia or known type III hyperlipoproteinemia (familial dysbetalipoproteinemia).
* Has fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain.
* Has uncontrolled hypertension
* Has had inflammatory bowel disease or any other malabsorption syndrome, or has had gastric bypass or any other surgical procedure for weight loss.
* Has a history of drug abuse or a history of high alcohol intake within the previous 2 years.
* Has type 1 or 2 diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in fasting plasma Low Density Lipoprotein cholesterol | Week 12 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in Triglycerides | Week 12 or Final Visit
Change from Baseline in Total Cholesterol | Week 12 or Final Visit
Change from Baseline in High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in Very Low Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in apolipoprotein A1 | Week 12 or Final Visit
Change from Baseline in apolipoprotein B | Week 12 or Final Visit
Change from Baseline in non- High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of Low Density Lipoprotein cholesterol/High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of Total Cholesterol/High Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of apolipoprotein A1/apolipoprotein B | Week 12 or Final Visit
Change from Baseline in high-sensitivity C-reactive protein | Week 12 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 1.81 mmol/L (70 mg/dL) | Week 12 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 2.59 mmol/L (100 mg/dL) | Week 12 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 3.37 mmol/L (130 mg/dL) | Week 12 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (86):
- United States (86):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Tuscaloosa, Alabama
  - Chandler, Arizona
  - Gilbert, Arizona
  - Glendale, Arizona
  - Tucson, Arizona
  - Artesia, California
  - Long Beach, California
  - Santa Ana, California
  - Santa Rosa, California
  - Tustin, California
  - Walnut Creek, California
  - Colorado Springs, Colorado
  - Golden, Colorado
  - Washington D.C., District of Columbia
  - Coral Gables, Florida
  - Fort Meyers, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Pembroke Pines, Florida
  - Pensacola, Florida
  - Pinellas Park, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Dunwoody, Georgia
  - Idaho Falls, Idaho
  - Aurora, Illinois
  - Chicago, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Overland Park, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - CantonAuburn, Maine
  - Scarborough, Maine
  - Baltimore, Maryland
  - Haverhill, Massachusetts
  - Ann Arbor, Michigan
  - Brooklyn Center, Minnesota
  - Edina, Minnesota
  - Olive Branch, Mississippi
  - St Louis, Missouri
  - Billings, Montana
  - Margate City, New Jersey
  - Wilwood, New Jersey
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Kettering, Ohio
  - Mentor, Ohio
  - Zanesville, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Altoona, Pennsylvania
  - Dowington, Pennsylvania
  - Sellerville, Pennsylvania
  - Warwick, Rhode Island
  - Goose Creek, South Carolina
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Irving, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burke, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Wauwatosa, Wisconsin